CLINICAL TRIAL: NCT03714750
Title: Treatment of Coronary Bifurcation Lesions: a Non-inferiority, Randomized, Controlled Procedural Outcomes Trial Comparing Reverse T and Protrusion Versus Double-kissing and Crush Stenting
Brief Title: Treatment of Coronary Bifurcation Lesions: Comparing Reverse T and Protrusion Versus Double-kissing and Crush Stenting
Acronym: TIPTAP-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tommaso Gori (Other)
Responsible Party: Sponsor-Investigator, Tommaso Gori, Prof. Dr. Tommaso Gori, PhD, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIP TAP I
Record Dates: First submitted 2018-10-04; First posted 2018-10-22 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease
Keywords: bifurcation coronary lesions; interventional technique of coronary lesions; Double kissing and crush; DK crush; Reverse TAP; reverse T-and-protrusion
MeSH Terms: conditions — Coronary Artery Disease; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DK crush (Active Comparator): Percutaneous revascularization of true coronary bifurcation stenosis (Medina 1,1,1 or 0,1,1) with double kissing and crush technique
  Interventions: Procedure: DK crush
- Reverse TAP (Experimental): Percutaneous revascularization of true coronary bifurcation Stenosis (Medina 1,1,1 or 0,1,1) with reverse T and protrusion technique
  Interventions: Procedure: Reverse TAP

INTERVENTIONS:
Procedure: DK crush — revascularization of true coronary bifurcation stenosis in DK crush technique
  Arms: DK crush
Procedure: Reverse TAP — revascularization of true coronary bifurcation stenosis in Reverse TAP technique
  Arms: Reverse TAP

SUMMARY:
Treatment of bifurcation coronary lesions may be challenging, and the best technique to be used in these settings remains to be established. While a single stent strategy is simpler and has been often encouraged, a number of studies show that the use of modern stent implantation techniques may bring some advantages in terms of target lesion failure during longer follow-up. Further, single-stent procedures are not possible at all in some settings, for instance when both main and side branch have similar diameters and present both relevant disease, particularly when the angle between the vessels is lower than 70°. Recent randomized data demonstrate the superiority of the technique called double kissing and crush (DK-Crush) over provisional stenting in this setting. The DK-Crush technique is however cumbersome, time-consuming and requires very experienced operators. The investigators therefore plan to undertake a randomized study comparing a novel interventional technique against DK-crush in the setting of true bifurcation lesions (Medina lesions type 1,1,1 or 0,1,1).

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the inclusion criteria:

* Documented heart team (as per guidelines) decision for revascularization via PCI
* Planned percutaneous coronary intervention (PCI) for a bifurcation stenosis with both branches >2.5mm and with a stenosis >50% and clinical indication to percutaneous intervention, including:

  * Ischemic symptoms, OR
  * Positive non-invasive imaging for ischemia, OR
  * Positive Flow Fractional Reserve (FFR), OR
  * mean lumen area (MLA) <6mm^2 for the left main or <4mm^2 for epicardial vessels as assessed by intracoronary imaging (IVUS, OCT)
* Vessel diameter ≤5.00mm
* True bifurcation lesion type 1,1,1 or 0,1,1
* Patient ≥18 years old

Exclusion Criteria:

* Cardiogenic shock
* Trifurcation if all vessels are ≥2.75mm diameter
* Either bifurcation vessel not suitable for stenting
* History of stenting in target bifurcation lesion
* Participation in another investigational drug or device study
* Patient unable to give informed consent
* Women of child-bearing potential or lactating
* In-stent restenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Stent Expansion in the side branch (defined as the vessel which received the first stent) | through study completion, an average of 2 hours
  Ratio of the minimum stent area of the side branch and the maximum stent area of the side branch

SECONDARY OUTCOMES:
fluoroscopy time | through study completion, an average of 2 hours
  Time of radiation during intervention
procedural time | through study completion, an average of 2 hours
  time of procedure ("Skin-to-Skin"-time)
use of coronary wires | through study completion, an average of 2 hours
  amount of coronary wires used during procedure
protocol success | through study completion, an average of 2 hours
  the Intervention is performed according to the protocol (including final kissing PTCA)
Min. lumen Diameter in main branch | through study completion, an average of 2 hours
  Minimum lumen Diameter in the main branch
Percentage of Stenosis in main branch | through study completion, an average of 2 hours
  Percentage of Stenosis in the main branch
Min. lumen Diameter in side branch | through study completion, an average of 2 hours
  Minimum lumen Diameter in the side branch
Percentage of Stenosis in side branch | through study completion, an average of 2 hours
  Percentage of Stenosis in the side branch
Procedural success | through study completion, an average of 2 days
  procedural success defined by angiographic success (no residual Stenosis of more than 20% at the end of Radiation) AND no periprocedural complications (including STEMI, new Q-wave myocardial infarction (MI), death, stent thrombosis, by-pass surgery, peri-procedural cardiac biomarker release according to the third universal definition of myocardial infarction) at discharge

OTHER OUTCOMES:
average stent eccentricity index (SEI) in the side branch | through study completion, an average of 2 hours
  optical coherence tomography endpoint, calculated as the Ratio of the Minimum to Maximum stent Diameter in the side branch
average stent eccentricity index (SEI) in the main branch | through study completion, an average of 2 hours
  optical coherence tomography endpoint, calculated as the Ratio of the Minimum to Maximum stent Diameter in the main branch
Minimum lumen diameter in the main branch | through study completion, an average of 2 hours
  optical coherence tomography endpoint, Minimum lumen Diameter in the main branch
Mean lumen diameter in the main branch | through study completion, an average of 2 hours
  optical coherence tomography endpoint, Mean lumen Diameter in the main branch
Minimum lumen area in the main branch | through study completion, an average of 2 hours
  optical coherence tomography endpoint, Minimum lumen Area in the main branch
Mean lumen area in the main branch | through study completion, an average of 2 hours
  optical coherence tomography endpoint, Mean lumen Area in the main branch
Minimum lumen diameter in the side branch | through study completion, an average of 2 hours
  optical coherence tomography endpoint, Minimum lumen Diameter in the side branch
Mean lumen diameter in the side branch | through study completion, an average of 2 hours
  optical coherence tomography endpoint, Mean lumen Diameter in the side branch
Minimum lumen area in the side branch | through study completion, an average of 2 hours
  optical coherence tomography endpoint, Minimum lumen area in the side branch
Mean lumen area in the side branch | through study completion, an average of 2 hours
  optical coherence tomography endpoint, Mean lumen Area in the side branch
Side branch obstruction | through study completion, an average of 2 hours
  optical coherence tomography endpoint, side branch obstruction through malapposed struts expressed as mean ratio between maximum inter-strut opening and side branch ostium diameter
Strut malapposition at bifurcation | through study completion, an average of 2 hours
  optical coherence tomography endpoint, % struts malapposed

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Gori, Prof Dr, PhD, Principal Investigator — Center of Cardiology, Cardiology I, University hospital Mainz
Locations (1):
- Center of Cardiology, Cardiology I, university hospital Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abouelnour AE, Olschewski M, Makmur G, Ullrich H, Knorr M, Ahoopai M, Munzel T, Gori T. Six-months clinical and intracoronary imaging follow-up after reverse T and protrusion or double-kissing and crush stenting for the treatment of complex left main bifurcation lesions. Front Cardiovasc Med. 2023 Apr 27;10:1153652. doi: 10.3389/fcvm.2023.1153652. eCollection 2023. PMID 37180808
- [Derived] Olschewski M, Ullrich H, Knorr M, Makmur G, Ahoopai M, Munzel T, Gori T. Randomized non-inferiority TrIal comParing reverse T And Protrusion versus double-kissing and crush Stenting for the treatment of complex left main bifurcation lesions. Clin Res Cardiol. 2022 Jul;111(7):750-760. doi: 10.1007/s00392-021-01972-2. Epub 2021 Nov 24. PMID 34816311
- [Derived] Rakhimov K, Buono A, Anadol R, Ullrich H, Knorr M, Ahoopai M, Munzel T, Gori T. Randomised, non-inferiority, controlled procedural outcomes TrIal comParing reverse T And Protrusion versus double-kissing and crush stenting: protocol of the TIP TAP I randomised trial. BMJ Open. 2020 Jun 16;10(6):e034264. doi: 10.1136/bmjopen-2019-034264. PMID 32554736